CLINICAL TRIAL: NCT04995809
Title: Investigating the Effect of Pelvic Radiotherapy on the Intestinal Microbiome and Metabolome to Improve the Detection and Management of Gastrointestinal (GI) Toxicity.
Brief Title: Effect of Pelvic Radiotherapy on the Intestinal Microbiome and Metabolome
Acronym: EPRIMM
Status: Completed | Type: Observational
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: University of Liverpool (Other); University of Manchester (Other); Wythenshawe Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 21_DOG13_32
Record Dates: First submitted 2021-05-26; First posted 2021-08-09 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2024-10

CONDITIONS: Urinary Bladder Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms
Keywords: Pelvic radiotherapy; Microbiota; Metabolome; Gastrointestinal toxicity
MeSH Terms: conditions — Urinary Bladder Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EPRIMM study participants: No intervention: Questionnaires, food diaries and stool sample.

SUMMARY:
Eight in ten patients will develop bowel problems during radiotherapy, eg diarrhoea, pain and incontinence, half will develop difficult long-term bowel problems. It is not known why some people get bowel problems and others do not and there is no test to predict who will develop bowel problems following their treatment.

There is a link between the changes in the number and type of gut bacteria (the microbiome) in some bowel conditions and it is possible to test for these different bacteria in a simple stool sample using genetic testing. Also gut bacteria produce different gases in the stool called "volatile organic compounds" (VOCs), which can be measured in stool samples. Specific VOC patterns have been seen in other bowel conditions and small studies suggesting that there are specific VOC and gut bacteria patterns in the stool of those undergoing pelvic radiotherapy which may help to identify people who will get difficult bowel problems. Diet can change the microbiome/VOCs so diet change could improve bowel symptoms after radiotherapy.

The investigators would like to test stool samples of patients with womb, cervix or bladder cancer having pelvic radiotherapy to see if there are differences in the number/type of gut bacteria and VOCs between those who get severe bowel symptoms compared to those with mild bowel symptoms. They also want to see whether these differences in VOCs or gut bacteria can tell who will develop severe bowel symptoms during or after radiotherapy and determine the effect of diet.

The first step is to run the study on a small scale to confirm that a larger study would work. This will make sure the investigators can recruit and consent people safely and will test the best ways of measuring bowels symptoms using several questionnaire options. They will collect the information needed to work out how many people would be needed in a large trial to fully test the theory. Ultimately, the investigators would like to use differences in the number/type of gut bacteria and VOCs to find ways to better prevent and treat bowel problems after pelvic radiotherapy.

DETAILED DESCRIPTION:
Background 80% of patients develop GI-toxicity during pelvic radiotherapy and half develop chronic GI-toxicity. This manifests as diarrhoea, pain, bleeding and incontinence. Unlike many diseases, the triggering event, i.e. radiotherapy, is known, enabling the identification of specific pathophysiological changes. The metabolomic and microbiomic profile of patients undergoing pelvic radiotherapy and the link with GI-toxicity has not been fully explored. Studies suggest radiation alters the gut microbiome, altering microbial diversity. Higher pre-radiotherapy diversity has been seen in those with no GI symptoms with reducing diversity as GI-toxicity increases and an association between low microbial diversity and severity of chronic GI-toxicity. Dietary change can alter microbial composition. Faecal VOCs are chemicals that exist in the gaseous phase at ambient temperature and form the faecal metabolome, the result of the interaction between the gut microbiota and cell metabolism. VOCs can be identified using established techniques and unique VOCs patterns have been identified in specific GI diseases. Early data suggest differences in VOCs between patients with high vs low levels of GI-toxicity. Metabolomic and microbiomic profiling and manipulation has the potential to advance understanding of disease-related pathways to predict, prevent and treat GI-toxicity.

Rationale GI-toxicity is a significant cause of morbidity both during and after pelvic radiotherapy to the extent that it adversely affects quality of life. There is a paucity of research into this condition. The metabolomic and microbiomic profile of patients undergoing pelvic radiotherapy and the link with GI-toxicity has not been fully explored. Studies suggest radiation alters the gut microbiome, altering microbial diversity. Higher pre-radiotherapy diversity has been seen in those with no GI symptoms with reducing diversity as GI-toxicity increases and an association between low microbial diversity and severity of chronic GI-toxicity. Dietary change can alter microbial composition. Unique VOCs patterns have been identified in specific GI diseases. Early data suggest differences in VOCs between patients with high vs low levels of GI-toxicity. Metabolomic and microbiomic profiling and manipulation has the potential to advance understanding of disease-related pathways to predict, prevent and treat GI-toxicity.

By comparing samples collected pre and post radiotherapy the investigators aim to identify potential biomarkers. They are going to integrate metadata indicating a negative GI response to the therapy, i.e. GI toxicity symptoms from validated questionnaires, with microbial community data and VOCs data in order to identify markers (VOCs or bacteria) that increase with symptoms. They will also identify which species make patients more susceptible to negative outcomes by analysing the community pre-treatment.

Previous literature using culture based methods showed an increase in E. coli and Staphylococcus spp. and the investigators will determine whether they can confirm this. In terms of VOCs, they will look for markers of inflammation, e.g. aldehydes. It has been proposed that there are similarities between radiation-induced GI-toxicity and IBD, particularly Crohn's disease, therefore it would be interesting to see whether there is a similar dysbiosis of the microbial community and VOCs profile to that observed in Crohn's disease, i.e. whether decreased species diversity, increased Bacteroides species and Enterobacteriaceae coupled with a decrease in Faecal bacterium are also observed in patients with severe GI toxicity symptoms.

Potential interventions to modify the gut microbiome, e.g. diet, pre/probiotics, synthetic faecal microbiota transplantation, are in wide clinical research use currently in other related clinical areas, e.g. inflammatory bowel disease, and would be the types of interventions that may be indicated by information from this work and the subsequent definitive study.

The objectives of the subsequent definitive study are as follows:

1. Determine the differences in VOC profile/microbiome in patients with the most severe vs least severe GI-toxicity at 4 weeks and 6 months.
2. Determine the differences in VOC profile/microbiome at baseline in patients who develop the most severe vs least severe GI-toxicity at 4 weeks and 6 months.
3. Characterise disease-related pathways for GI-toxicity to identify potential therapeutic targets, including dietary.

ELIGIBILITY:
Inclusion Criteria:

* Pelvic radiotherapy-cervix/endometrial/bladder cancer.
* ≥18 years.
* Able to consent.
* Able to complete questionnaires.

Exclusion Criteria:

* Pre-existing GI disease
* Abdominopelvic surgery within preceding 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients will be identified from new patient referrals to oncology clinics for pelvic radiotherapy to treat cervix, endometrial or bladder cancer
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2023-07-21 (Actual)

PRIMARY OUTCOMES:
Rate of recruitment | 12 months
  Recruitment rates: can we achieve sufficient recruitment to the study? Are patients willing to participate?
Acceptability of recruitment | 12 months
  Acceptability of recruitment process to patient cohort measured using internally generated non-validated questionnaire led by the research nurse
Patient experience of study | 6 months
  Experience of the study process by patient cohort measured using internally generated non-validated questionnaire led by the research nurse
Stool sample collection | 6 months
  Practicality and acceptability of obtaining stool samples for patient cohort measured using internally generated non-validated questionnaire led by the research nurse
Attrition rates | 18 months
  Rate of patient leaving the study before completing
Reason for attrition | 18 months
  Reason for patient leaving the study before completing

SECONDARY OUTCOMES:
Acceptability of questionnaires/food diaries | 6 months
  Acceptability of questionnaires and food diaries to patient cohort measured using internally generated non-validated questionnaire led by the research nurse
Completion of information | 6 months
  Proportion of patients who complete the study eg rate of attrition of patients and rate of missing data items
The number of participants required to take part in a larger multicentre trial which will identify microbiome/VOC profiles which confer risk of GI toxicity | 24 months
  To identify microbiome (diversity or composition) or VOCs profile that confers risk of GI-toxicity and that is associated with participants greater severity of GI-toxicity in response in response to radiotherapy in the acute and chronic phases
The number of participants required to take part in a larger multicentre trial which will identify potential therapeutic targets from metabolomic and microbiomic profiling | 24 months
  To use metabolomic and microbiomic profiling to further understand the pathophysiology of GI-toxicity to identify potential therapeutic targets for treatment and/or prevention, including dietary targets

OTHER OUTCOMES:
Microbiome data (DNA reads) | 24 months
  Obtain initial data regarding microbiome (diversity or composition) associated with risk of GI-toxicity and that is associated with greater severity of GI-toxicity in response in response to radiotherapy in the acute and chronic phases
VOC profile by solid-phase microextraction followed by gas chromatography-mass spectrometry SPME-GC/MS | 24 months
  Obtain initial data (peak area/metabolite(VOC)/sample) regarding VOCs profile associated with risk of GI-toxicity and that is associated with greater severity of GI-toxicity in response in response to radiotherapy in the acute and chronic phases.
Metabolomic profiling by SPME-GC/MS | 24 months
  To use metabolomic profiling to further understand the pathophysiology of GI-toxicity to identify potential therapeutic targets for treatment and/or prevention, including dietary targets
Microbiomic profiling by bacterial 16S rRNA metabarcoding sequencing | 24 months
  To use microbiomic profiling ( data table containing number of reads/species/sample) to further understand the pathophysiology of GI-toxicity to identify potential therapeutic targets for treatment and/or prevention, including dietary targets

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Henson, MBBS PhD, Principal Investigator — The Christie NHS Foundation Trust
Locations (1):
- Louise James, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wedlake L, Thomas K, McGough C, Andreyev HJ. Small bowel bacterial overgrowth and lactose intolerance during radical pelvic radiotherapy: An observational study. Eur J Cancer. 2008 Oct;44(15):2212-7. doi: 10.1016/j.ejca.2008.07.018. Epub 2008 Aug 27. PMID 18760593
- [Background] Andreyev J. Gastrointestinal symptoms after pelvic radiotherapy: a new understanding to improve management of symptomatic patients. Lancet Oncol. 2007 Nov;8(11):1007-17. doi: 10.1016/S1470-2045(07)70341-8. PMID 17976611
- [Background] Gami B, Harrington K, Blake P, Dearnaley D, Tait D, Davies J, Norman AR, Andreyev HJ. How patients manage gastrointestinal symptoms after pelvic radiotherapy. Aliment Pharmacol Ther. 2003 Nov 15;18(10):987-94. doi: 10.1046/j.1365-2036.2003.01760.x. PMID 14616164
- [Background] Nam YD, Kim HJ, Seo JG, Kang SW, Bae JW. Impact of pelvic radiotherapy on gut microbiota of gynecological cancer patients revealed by massive pyrosequencing. PLoS One. 2013 Dec 18;8(12):e82659. doi: 10.1371/journal.pone.0082659. eCollection 2013. PMID 24367534
- [Background] Lam V, Moulder JE, Salzman NH, Dubinsky EA, Andersen GL, Baker JE. Intestinal microbiota as novel biomarkers of prior radiation exposure. Radiat Res. 2012 May;177(5):573-83. doi: 10.1667/rr2691.1. Epub 2012 Mar 23. PMID 22439602
- [Background] Kim YS, Kim J, Park SJ. High-throughput 16S rRNA gene sequencing reveals alterations of mouse intestinal microbiota after radiotherapy. Anaerobe. 2015 Jun;33:1-7. doi: 10.1016/j.anaerobe.2015.01.004. Epub 2015 Jan 16. PMID 25600706
- [Background] Manichanh C, Varela E, Martinez C, Antolin M, Llopis M, Dore J, Giralt J, Guarner F, Malagelada JR. The gut microbiota predispose to the pathophysiology of acute postradiotherapy diarrhea. Am J Gastroenterol. 2008 Jul;103(7):1754-61. doi: 10.1111/j.1572-0241.2008.01868.x. Epub 2008 Jun 28. PMID 18564125
- [Background] Goudarzi M, Mak TD, Jacobs JP, Moon BH, Strawn SJ, Braun J, Brenner DJ, Fornace AJ Jr, Li HH. An Integrated Multi-Omic Approach to Assess Radiation Injury on the Host-Microbiome Axis. Radiat Res. 2016 Sep;186(3):219-34. doi: 10.1667/RR14306.1. Epub 2016 Aug 11. PMID 27512828
- [Background] Wang A, Ling Z, Yang Z, Kiela PR, Wang T, Wang C, Cao L, Geng F, Shen M, Ran X, Su Y, Cheng T, Wang J. Gut microbial dysbiosis may predict diarrhea and fatigue in patients undergoing pelvic cancer radiotherapy: a pilot study. PLoS One. 2015 May 8;10(5):e0126312. doi: 10.1371/journal.pone.0126312. eCollection 2015. PMID 25955845
- [Background] Reis Ferreira M, Andreyev HJN, Mohammed K, Truelove L, Gowan SM, Li J, Gulliford SL, Marchesi JR, Dearnaley DP. Microbiota- and Radiotherapy-Induced Gastrointestinal Side-Effects (MARS) Study: A Large Pilot Study of the Microbiome in Acute and Late-Radiation Enteropathy. Clin Cancer Res. 2019 Nov 1;25(21):6487-6500. doi: 10.1158/1078-0432.CCR-19-0960. Epub 2019 Jul 25. PMID 31345839
- [Background] Cui M, Xiao H, Li Y, Zhou L, Zhao S, Luo D, Zheng Q, Dong J, Zhao Y, Zhang X, Zhang J, Lu L, Wang H, Fan S. Faecal microbiota transplantation protects against radiation-induced toxicity. EMBO Mol Med. 2017 Apr;9(4):448-461. doi: 10.15252/emmm.201606932. PMID 28242755
- [Background] David LA, Maurice CF, Carmody RN, Gootenberg DB, Button JE, Wolfe BE, Ling AV, Devlin AS, Varma Y, Fischbach MA, Biddinger SB, Dutton RJ, Turnbaugh PJ. Diet rapidly and reproducibly alters the human gut microbiome. Nature. 2014 Jan 23;505(7484):559-63. doi: 10.1038/nature12820. Epub 2013 Dec 11. PMID 24336217
- [Background] Reade S, Mayor A, Aggio R, Khalid T, Pritchard DM, Ewer AK, et al. Optimisation of Sample Preparation for Direct SPME-GC-MS Analysis of Murine and Human Faecal Volatile Organic Compounds for Metabolomic Studies. J Anal Bioanal Tech. 2014;5(2).
- [Background] Xu X, Xu P, Ma C, Tang J, Zhang X. Gut microbiota, host health, and polysaccharides. Biotechnol Adv. 2013 Mar-Apr;31(2):318-37. doi: 10.1016/j.biotechadv.2012.12.009. Epub 2012 Dec 30. PMID 23280014
- [Background] Hough R, Archer D, Probert C. A comparison of sample preparation methods for extracting volatile organic compounds (VOCs) from equine faeces using HS-SPME. Metabolomics. 2018;14(2):19. doi: 10.1007/s11306-017-1315-7. Epub 2018 Jan 4. PMID 29367839
- [Background] Mikami T, Aoki M, Kimura T. The application of mass spectrometry to proteomics and metabolomics in biomarker discovery and drug development. Curr Mol Pharmacol. 2012 Jun;5(2):301-16. doi: 10.2174/1874467211205020301. PMID 22122469
- [Background] Probert CS. Role of faecal gas analysis for the diagnosis of IBD. Biochem Soc Trans. 2011 Aug;39(4):1079-80. doi: 10.1042/BST0391079. PMID 21787351
- [Background] Probert CS, Ahmed I, Khalid T, Johnson E, Smith S, Ratcliffe N. Volatile organic compounds as diagnostic biomarkers in gastrointestinal and liver diseases. J Gastrointestin Liver Dis. 2009 Sep;18(3):337-43. PMID 19795029
- [Background] Probert CS, Jones PR, Ratcliffe NM. A novel method for rapidly diagnosing the causes of diarrhoea. Gut. 2004 Jan;53(1):58-61. doi: 10.1136/gut.53.1.58. PMID 14684577
- [Background] Covington JA, Wedlake L, Andreyev J, Ouaret N, Thomas MG, Nwokolo CU, Bardhan KD, Arasaradnam RP. The detection of patients at risk of gastrointestinal toxicity during pelvic radiotherapy by electronic nose and FAIMS: a pilot study. Sensors (Basel). 2012 Sep 26;12(10):13002-18. doi: 10.3390/s121013002. PMID 23201982
- [Background] Sokol H, Adolph TE. The microbiota: an underestimated actor in radiation-induced lesions? Gut. 2018 Jan;67(1):1-2. doi: 10.1136/gutjnl-2017-314279. Epub 2017 May 4. No abstract available. PMID 28473631
- [Background] Stringer AM, Al-Dasooqi N, Bowen JM, Tan TH, Radzuan M, Logan RM, Mayo B, Keefe DM, Gibson RJ. Biomarkers of chemotherapy-induced diarrhoea: a clinical study of intestinal microbiome alterations, inflammation and circulating matrix metalloproteinases. Support Care Cancer. 2013 Jul;21(7):1843-52. doi: 10.1007/s00520-013-1741-7. Epub 2013 Feb 10. PMID 23397098
- [Background] Ferreira MR, Muls A, Dearnaley DP, Andreyev HJ. Microbiota and radiation-induced bowel toxicity: lessons from inflammatory bowel disease for the radiation oncologist. Lancet Oncol. 2014 Mar;15(3):e139-47. doi: 10.1016/S1470-2045(13)70504-7. PMID 24599929
- See also: Lay summary of EPRIMM results — https://www.hra.nhs.uk/planning-and-improving-research/application-summaries/research-summaries/eprimm/